CLINICAL TRIAL: NCT02481791
Title: Study to Evaluate the Optimal Dose of Remifentanil Required to Ensure Apnoea During Magnetic Resonance Imaging of the Heart Under General Anaesthesia
Brief Title: Study to Evaluate the Optimal Dose of Remifentanil During MRI of the Heart Under General Anaesthesia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 146613
Record Dates: First submitted 2015-06-19; First posted 2015-06-25 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Children; Heart Diseases; Anaesthesia; Magnetic Resonance Imaging
MeSH Terms: conditions — Heart Diseases | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remifentanil (Experimental): Induction Phase: A dose of remifentanil 1mcg/kg by slow bolus, will be given to facilitate endotracheal intubation. Further doses of either remifentanil (0.5 mcg/kg) or propofol (1-2mg/kg) may be given to ensure an anaesthetised patient.
  Settling Period: An infusion of the test dose of remifentanil will be commenced from an infusion prepared prior to the patient being anaesthetised. 1mg of Remifentanil (one vial) will be diluted to a volume of 50mls in normal saline 0.9% in a 50ml syringe. Maintenance dose of propofol 130 mcg/Kg/min for the first 5 minutes reduced to 100 mcg/kg/min thereafter. 40mls of propofol 1% (10mg/ml) will be drawn undiluted into a 50ml syringe. During the settling period further doses of either remifentanil (0.5 mcg/kg) or propofol (1-2mg/kg) may be given.
  Equilibrium Period: During this period propofol will be infused at a constant rate of 100mcg/kg/min.
  Interventions: Drug: Remifentanil and/or propofol; Drug: propofol

INTERVENTIONS:
Drug: Remifentanil and/or propofol — Induction Phase: A dose of remifentanil 1mcg/kg by slow bolus, will be given to facilitate endotracheal intubation. Further doses of either remifentanil (0.5 mcg/kg) or propofol (1-2mg/kg) may be given to ensure an anaesthetised patient.
Drug: Remifentanil and/or propofol — Settling Period: An infusion of the test dose of remifentanil will be commenced from an infusion prepared prior to the patient being anaesthetised. 1mg of Remifentanil (one vial) will be diluted to a volume of 50mls in normal saline 0.9% in a 50ml syringe. Maintenance dose of propofol 130 mcg/Kg/min for the first 5 minutes reduced to 100 mcg/kg/min thereafter. 40mls of propofol 1% (10mg/ml) will be drawn undiluted into a 50ml syringe. During the settling period further doses of either remifentanil (0.5 mcg/kg) or propofol (1-2mg/kg) may be given.
Drug: propofol — Equilibrium Period: During this period propofol will be infused at a constant rate of 100mcg/kg/min

SUMMARY:
What is the optimal maintenance dose of remifentanil to ensure apnoea, during breath hold episodes in children having cardiac MR imaging with general anaesthesia?

DETAILED DESCRIPTION:
The management of congenital heart disease depends upon accurate imaging of the heart to define anatomical abnormalities. The use of magnetic resonance imaging has grown in response to this need. Young children, however, are unable to cooperate sufficiently to allow the scan to occur; this necessitates the use of general anaesthesia.

The optimal anaesthetic management of children in this situation is complex. Imaging of an acceptable quality depends on a low (normal) heart rate which is relatively constant during the scan and frequent breath holds to avoid respiratory artefacts. Children undergoing such scans commonly have significant cardiac and non-cardiac disease. A technique, currently used at Alder Hey Hospital, is to use intravenous agents to provide anaesthesia: commonly a mixture of the intravenous anaesthetic propofol and the potent opiate remifentanil. The patient's own ventilation is suppressed by the use of remifentanil which also reduces heart rate and heart rate variability. Controlled ventilation is provided via a ventilator and endotracheal tube. Adequate doses of remifentanil are required to ensure suppression of the patient's ventilation whilst excess doses are avoided to reduce the risk of adverse effects (primarily arterial hypotension) and ensure rapid recovery.

Remifentanil dose has been studied during surgery(3-6), however this is a unique indication and optimal dosage has not been formally studied. In particular the absence of any stimulation from surgery is likely to mean that substantially lower doses of remifentanil will be required.

ELIGIBILITY:
Inclusion Criteria:

* Children of one year (of age) or older and younger than 7 years of age.
* Scheduled for cardiac MR imaging under general anaesthesia at Alder Hey Children's Hospital.
* Parental Consent

Exclusion Criteria:

* Hypersensitivity to any study drug
* Known abnormal response to opiate analgesics or co-morbidity associated with abnormal central control of breathing
* Families unable to understand or complete consent
* Any other contraindication to proposed anaesthetic technique: at the discretion of the responsible anaesthetist.
* Documented significant renal or hepatic dysfunction

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Diaphragm movement | 30 seconds
  The primary outcome will be movement of the diaphragm during the single test apnoea. The dose of remifentanil will be judged:
  * A success. If no movement of the diaphragm is detected by MRI imaging during a 30 second test apnoea.
  * A failure. If movement of the diaphragm is detected during the test apnoea.

SECONDARY OUTCOMES:
Scan Quality | 1 hour
  • quality of the scan from the respiratory gated sequence (graded by the radiologist who will be blinded to the dose)
Heart Rate | 1 hour
  • highest and lowest heart rate (during equilibrium and study period)
Blood pressure | 1 hour
  • lowest blood pressure (during equilibrium and study period)
Emergence time | 1 hour
  • time to emergence (waking up) at end of scan

CONTACTS AND LOCATIONS:
Locations (1):
- Alder Hey Children's Hospital, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Background] Syed SK, Corry P. Cardiac Imaging under general anaesthesia for children with congenital heart disease. Our experience. Abstract presentation, APAGBI scientific meeting. 2012.
- [Background] Chanavaz C, Tirel O, Wodey E, Bansard JY, Senhadji L, Robert JC, Ecoffey C. Haemodynamic effects of remifentanil in children with and without intravenous atropine. An echocardiographic study. Br J Anaesth. 2005 Jan;94(1):74-9. doi: 10.1093/bja/aeh293. Epub 2004 Oct 14. PMID 15486003
- [Background] Crawford MW, Hayes J, Tan JM. Dose-response of remifentanil for tracheal intubation in infants. Anesth Analg. 2005 Jun;100(6):1599-1604. doi: 10.1213/01.ANE.0000150940.57369.B5. PMID 15920180
- [Background] Hume-Smith H, McCormack J, Montgomery C, Brant R, Malherbe S, Mehta D, Ansermino JM. The effect of age on the dose of remifentanil for tracheal intubation in infants and children. Paediatr Anaesth. 2010 Jan;20(1):19-27. doi: 10.1111/j.1460-9592.2009.03190.x. Epub 2009 Nov 23. PMID 19968808
- [Background] Min SK, Kwak YL, Park SY, Kim JS, Kim JY. The optimal dose of remifentanil for intubation during sevoflurane induction without neuromuscular blockade in children. Anaesthesia. 2007 May;62(5):446-50. doi: 10.1111/j.1365-2044.2007.05037.x. PMID 17448054
- [Background] Ross AK, Davis PJ, Dear Gd GL, Ginsberg B, McGowan FX, Stiller RD, Henson LG, Huffman C, Muir KT. Pharmacokinetics of remifentanil in anesthetized pediatric patients undergoing elective surgery or diagnostic procedures. Anesth Analg. 2001 Dec;93(6):1393-401, table of contents. doi: 10.1097/00000539-200112000-00008. PMID 11726413
- [Background] Whitehead J, Brunier H. Bayesian decision procedures for dose determining experiments. Stat Med. 1995 May 15-30;14(9-10):885-93; discussion 895-9. doi: 10.1002/sim.4780140904. PMID 7569508
- [Background] Whitehead J, Williamson D. Bayesian decision procedures based on logistic regression models for dose-finding studies. J Biopharm Stat. 1998 Jul;8(3):445-67. doi: 10.1080/10543409808835252. PMID 9741859
- [Background] Zhou Y, Whitehead J. Practical Implementation of Bayesian Dose-Escalation Procedures. Drug Information Journal. 2003;37(1):45-59.
- [Background] R Core Team R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. 2013.